CLINICAL TRIAL: NCT04874883
Title: Intestinal Function of Patients With Colon Neoplasia, Airways and Upper Digestives Subjected to Surgical Treatment: Impact of the Use of Symbiotics
Brief Title: Effect of the Use of Symbiotics in Patients With Colon Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Minas Gerais (Other)
Collaborators: Simone de Vasconcelos Generoso (Unknown); Luísa Martins Trindade (Unknown); Rodrigo Gomes Silva (Unknown); Maria Isabel Toulson Davisson Correia (Unknown)
Responsible Party: Principal Investigator, Maria Isabel Toulson Davisson Correia, Sponsor-Investigator, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 24375713.0.0000.5149
Record Dates: First submitted 2021-04-22; First posted 2021-05-06 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-04

CONDITIONS: Symbiotic; Cancer Colorectal; Cancer Head Neck; Intestinal Dysbiosis; Diarrhea; Intestinal Microbiota; Nutritional Status
MeSH Terms: conditions — Colonic Neoplasms; Head and Neck Neoplasms; Diarrhea | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The study will be double-masked and individuals will be randomly divided into two groups: Symbiotic group (S) - will receive the symbiotic (association of fructooligosaccharide, prebiotic, and four probiotic strains: Lactobacillus casei, Lactobacillus rhamnosus, Lactobacillus Acidophilus, and Bifidobacterium bifidum) enterally or orally in the amount of a sachet, twice a day. Control Group (C) will receive maltodextrin placebo (carbohydrate easily absorbed and digested, not fermented by colonic bacteria and which does not interfere in the microbial ecology of the gastrointestinal tract or in the metabolism and function of the intestine), either enterally or orally in a sachet. hours until hospital discharge.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All individuals directly involved in the research will be masked. The modules used in the study were masked by an individual external to the research, being the only one who knew the composition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Active Comparator): You will receive 6 grams of the symbiotic (association of fructooligosaccharides, prebiotics, and four probiotic strains: Lactobacillus casei, Lactobacillus rhamnosus, Lactobacillus Acidophilus, and Bifidobacterium bifidum) either enterally or twice a day.
  Interventions: Dietary Supplement: Simbyotic
- Control Group (Placebo Comparator): Will receive 6 grams of the maltodextrin placebo (carbohydrate easily absorbed and digested, not fermented by colonic bacteria and which does not interfere in the microbial ecology of the gastrointestinal tract or in the metabolism and function of the intestine), either enterally or orally in two sachets times a day
  Interventions: Device: Control Group

INTERVENTIONS:
Dietary Supplement: Simbyotic — 6 grams of the symbiotic will be administered twice a day
  Arms: Intervention Group
Device: Control Group — 6 grams of the maltodextrin will be administered twice a day
  Arms: Control Group

SUMMARY:
Due to the high incidence, cancer and the concomitant presence of malnutrition are currently a worldwide public health problem. The loss of weight and body tissues is a common condition in cancer patients with lesions of the airways and digestive tract and is related to anorexia and the presence and duration of gastrointestinal symptoms, such as diarrhea. The latter directly interferes with the progression of enteral diets, which are administered in order to provide adequate nutritional support for the recovery of patients and nutritional status. In this sense, the importance of measures to help reduce diarrhea episodes is reinforced, aiming at the adequate infusion of enteral diets and, consequently, nutritional needs. It is known that the use of antimicrobials is closely related to the increased incidence of nasocomial diarrhea, as it facilitates colonization by pathogenic bacteria, such as Clostridium difficile. In addition, nosocomial diarrhea is a very relevant occurrence due to the financial burden it causes for the hospital institution, which can also worsen the patient's clinical condition, since he is weakened due to the underlying disease. Despite these important aspects, studies carried out with the aim of reducing diarrhea episodes in patients with airway and digestive lesions are still not described in the literature. In this context, the use of symbiotics presents itself as a possibly beneficial alternative, considering the role of probiotics and prebiotics in the modulation of intestinal function. In this sense, this work aims to evaluate the impact of perioperative supplementation with symbiotic on clinical outcomes and intestinal function of patients with colon cancer and digestive airways undergoing colorectal resection. It is assumed that the use of symbiotics could have better results than the use of probiotics and isolated prebiotics.

DETAILED DESCRIPTION:
Most cancer patients have a compromised nutritional status, 80% are malnourished at the time of the initial diagnosis. It is known that in patients with airway and digestive cancer the risk of malnutrition is increased, due to changes caused by the location of the tumor such as dysphagia, odynophagia and changes in taste.

The clinical effects of malnutrition are manifested by difficulty in healing after surgery, increased risk of infection and treatment toxicity, in addition to greater demand for care and hospital costs. Therefore, it is of utmost importance to provide adequate nutritional needs to these patients, since adequate nutritional therapy (NT) is able to improve their clinical response and prognosis.

Nutritional support is seen as an important strategy for the treatment and recovery of these patients, since it promotes greater adequacy of nutritional support, improving nutritional status as well as response to treatment and immune function, in addition to improving quality of life and reducing hospital costs. However, gastrointestinal complications, such as diarrhea, represent important causes for not receiving the planned enteral diet volume, or the patient's intake inadequacy, which causes an insufficient supply of calories, proteins, vitamins and minerals over the days, contributing with worsening nutritional status, as well as increased hospital stay and costs with hospitalization.

Diarrhea affects about 16% to 63% of patients on enteral nutrition. The most frequent causes of diarrhea in cancer patients are related to medications, such as antibiotics, antacids with magnesium, lactulose, laxatives, supplements with potassium and phosphorus and medications with sorbitol6. Other possible causes of diarrhea include hypoalbuminemia, rapid infusion and intolerance to some component of the diet, infectious causes such as the presence of Clostridium difficile, severe malnutrition and, more rarely with the use of industrialized diets, bacterial contamination of the enteral formula.

In particular, the presence of nosocomial diarrhea - defined as infectious diarrhea acquired in a hospital environment - increases the length of stay of patients (eight days, on average), increases the likelihood of infections in surgical wounds, and consequently, hospital mortality. Among the identifiable causes of this type of diarrhea, the indiscriminate use of antimicrobials has been identified as an important predisposing factor, particularly in facilitating colonization and intestinal infection by Clostridium difficile. This bacterium has an incidence between 5% and 39%, with an increased incidence in hospitalized post-surgical patients.

Thus, it is necessary to study strategies that reduce the incidence of diarrhea in these patients. In this context, the use of probiotics and prebiotics seems to be an effective alternative, since the therapeutic effect in the treatment and prevention of intestinal diseases has been extensively researched.

Probiotics are live microorganisms that, when consumed in adequate and sufficient quantities, confer benefits to the health of the host. In addition, they compete with pathogenic bacteria for space and nutrients, blocking their effects and binding them to the intestinal mucosa. They produce antibacterial substances (bacteriocins), acidify the intestinal pH by fermentation and production of lactic acid, stimulate the production of mucin and increase the production and secretion of immunoglobulin A (sIgA). There is evidence that probiotics also contribute to the reduction of inflammatory mediators such as tumor necrosis factor (TNF) and growth transformation factor (TGF-β) that modulate the inflammatory response and favor immune balance. Lactobacillus casei, Lactobacillus rhamnosus, Lactobacillus acidophilus and Bifidobacterium are some of the probiotics that have benefits described in the literature.

Cimperman et al (2011), in a pilot study, double masked, controlled placebo evaluated the effect of treatment with probiotics in patients using antibiotics. The results showed that the administration of the probiotic Lactobacillus reuteri significantly reduced diarrhea compared to patients who received a placebo. Still, D'Souza et al (2002), Cremonini et al (2002) & McFarland (2006) concluded through meta-analyzes that the use of probiotics is associated with the prevention of diarrhea associated with the use of antibiotics in hospitalized patients.

Prebiotics are defined as food substances that, when ingested, are not digested and absorbed by the small intestine. When they reach the colon, they are used as a substrate for probiotics, selectively stimulating the growth of the intestinal microbiota in addition to producing short-chain fatty acids (SCFA) that are substrates for colonocytes. SCFAs also modulate the intestinal microbiota, maintain metabolism and promote a decrease in intestinal pH, thereby inhibiting the development of pathogenic microorganisms. Rushdi, Pichard & Khater (2004) evaluated in a prospective, double-masked controlled study the effect of adding soluble fiber to the enteral diet of patients hospitalized with diarrhea. Patients were randomly divided into two groups: control (enteral diet without soluble fiber) and treated (enteral diet with soluble fiber). The results showed a reduction in diarrhea episodes in the study patients, suggesting the prebiotic benefit of soluble fiber. Examples of prebiotics are fructooligosaccharides (FOS) and galactooligosaccharides (GOS).

These findings propose that interventions aimed at modulating intestinal function related to the prevention and control of diarrhea in cancer patients in the postoperative period deserve to be implemented and evaluated. However, these trials used different probiotic organisms, prebiotics, doses, duration of treatment and target audience, providing low reproducibility of the results. In addition, some studies have shown that symbiotics (defined as a combination of probiotics and prebiotics) can optimize the beneficial results in relation to the isolated use of probiotics in terms of modulating the immune system and the intestinal microbiota. It is suggested that under the action of symbiotics there will be better control of intestinal functioning and improved prognosis.

In this sense, evaluating the symbiotic administration in patients with colon, upper airway and digestive cancer undergoing surgical treatment would be a potentially beneficial alternative to be studied, since the consumption of this food component could lead to modulation of intestinal function, preventing diarrhea that, according to our data, occurs in 30% of the patients hospitalized at the Alfa Institute of Gastroenterology at UFMG.

General objective

To evaluate the impact of the symbiotic on the intestinal function of patients with malignant neoplasm of the colon, upper airways and digestive tract submitted to surgical treatment.

Specific objectives

* Assess the incidence of diarrhea in the study group;
* Identify other gastrointestinal symptoms such as stasis, vomiting, bloating;
* Identify and monitor the evolution of the nutritional status of patients through subjective global assessment, anthropometry and food consumption;
* Track postoperative complications, in general.

The study will be carried out at the Alfa Institute of Gastroenterology, Hospital das Clínicas, Federal University of Minas Gerais, located in Belo Horizonte, Minas Gerais.The sample will comprise 42 patients (21 in the intervention group and 21 in the control group). The sample calculation was performed according to Hulley et al. (2001), using the proportion of 30% improvement in the symptom of diarrhea with the use of symbiotic from the average of other studies, considering a range of 45% of the confidence interval (difference between the highest and the lowest value found) and 12% loss with the intervention, also observed in the reference studies. Individuals will be invited to participate in the study and will have a detailed explanation of the procedure and research in which they will be inserted, and must sign a free and informed consent form. Individuals who have inflammatory bowel diseases will be excluded; have previously undergone operations on the gastrointestinal tract; have used antibiotics, prebiotics, probiotics or symbiotics in the last 15 days and are using an enteral fiber diet. The study will be double-masked and the individuals will be randomly divided into two groups: Symbiotic group (S) - will receive the symbiotic (association of fructooligosaccharide, prebiotic, and four probiotic strains: Lactobacillus casei, Lactobacillus rhamnosus, Lactobacillus Acidophilus, and Bifidobacterium bifidum) enterally or orally in the amount of a sachet, twice a day. Control Group (C) will receive maltodextrin placebo (carbohydrate easily absorbed and digested, not fermented by colonic bacteria and which does not interfere in the microbial ecology of the gastrointestinal tract or in the metabolism and function of the intestine), either enterally or orally in a sachet. hours until hospital discharge. Personal information such as full name, medical record number, sex, age, marital status, origin, date of birth and hospitalization will be collected for patient identification. Information regarding the location of the tumor, type of tumor, age of diagnosis in years and months, type of previous and current treatment (surgical, radiotherapy and / or chemotherapy) use of antibiotics, comorbidities and presence or not of infection will be collected from the medical record . The evaluation of intestinal functioning will be made by direct questioning to patients and family members, as well as the nursing records. The occurrence or not of diarrhea (defined as more than three bowel movements / day), frequency and volume, whether or not gastrointestinal symptoms such as distension and abdominal pain during hospitalization will be assessed. Nutritional assessment will be carried out by Subjective Global Assessment proposed by Detsky (1987) and using anthropometric parameters: current weight, height, arm, tricipital skin fold, subscapular and biochemical.

The start of the diet in the postoperative period and the nutrient supply will be verified through the analysis of food consumption and / or infusion of the enteral diet, which was calculated according to the service protocol, contemplating 30 calories per kilogram of current weight.

Complications will be assessed through the daily assessment of the patient and medical records and classified according to the proposal by Dindo (2004).

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age, diagnosed with colorectal and head and neck cancer who will undergo a tumor resection operation

Exclusion Criteria:

* Individuals who have inflammatory bowel diseases will be excluded; have previously undergone operations on the gastrointestinal tract; have used antibiotics, prebiotics, probiotics or symbiotics in the last 15 days and are on an enteral fiber diet.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Diarrhea occurrence | Through study completion, an average of 2 years
  Assess the incidence of diarrhea by collecting information on the frequency and consistency of stools. Stool consistency will be classified using the Bristol scale.

SECONDARY OUTCOMES:
Nutritional status | Through study completion, an average of 2 years
  Monitor patients' nutritional status through subjective global assessment, weight, arm circumference, tricipital skinfold and food consumption.
Operative complications | Through study completion, an average of 2 years
  Evaluate operative complications, such as length of hospital stay, need for mechanical ventilation, need for enteral or parenteral nutritional therapy and mortality, through medical records

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Escola de Enfermagem - UFMG, Belo Horizonte, Minas Gerais
  - Ambulatório de Transplantes Hepáticos, Belo Horizonte, Minas Gerais

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Trindade LM, Borges AD, Carvalho RDO, Gomes BF, da Silva MT, Sette NSV, Rogerio L, Cavalcanti GG, Garcia APV, Cassali GD, Azevedo VA, Cardoso VN, Mauricio SF, Rodrigues LB, Valdes ST, da Silva RG, Generoso SV. Preoperative symbiotic supplementation modulates the intestinal microbiota of patients with colorectal cancer: Evidence from a randomized clinical trial. Nutrition. 2025 Dec 26;145:113080. doi: 10.1016/j.nut.2025.113080. Online ahead of print. PMID 41637916